CLINICAL TRIAL: NCT01686360
Title: Communicating Objective Risk for Personalized Decision Making About Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 816186
Record Dates: First submitted 2012-08-28; First posted 2012-09-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Control group 1: pre/post-test (No Intervention): Group receives pre and post test questions only.
- Control group 2: tool and pre/post-test (Experimental): Group receives decision tool without personalized information. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid
- Gail score in a percentage format (Experimental): Group receives Gail score in a percentage format. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid
- Gail score in a frequency format (Experimental): Group receives Gail score in a frequency format. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid
- Frequency + Average 50 year old (Experimental): Group receives Gail score in a frequency format as well as information about risk of breast cancer for the average 50 year old woman. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid
- Frequency + Mammography Data (Experimental): Group receives Gail score in a frequency format as well as information about the risks of mammography. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid
- Frequency + Mortality Data (Experimental): Group receives Gail score in a frequency format as well as information about mortality benefit of mammography. (Behavioral:Decision Aid)
  Interventions: Behavioral: Decision Aid
- Frequency + Avg 50 year old + Mamm Data + Mortality Data (Experimental): Group receives Gail score in a frequency format as well as information about breast cancer risk for the average 50 year old woman, information about the risks of mammography, risk of breast cancer for the average 50 year old woman, and information about the mortality benefit associated with mammography. (Behavioral: Decision Aid)
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid
  Arms: Control group 2: tool and pre/post-test; Frequency + Average 50 year old; Frequency + Avg 50 year old + Mamm Data + Mortality Data; Frequency + Mammography Data; Frequency + Mortality Data; Gail score in a frequency format; Gail score in a percentage format

SUMMARY:
The purpose of this study is to test the effects of objective risk information about breast cancer and mammography outcomes using a randomized control trial. Women between the ages of 35 and 49 will receive information about their personal risk for breast cancer and be randomly assigned to receive data about a woman who should be screened, data about the potential outcomes of screening, or data about breast cancer deaths. Two presentation formats will be tested and compared.

DETAILED DESCRIPTION:
This study will compare alternative strategies for the presentation of individualized information about the risks and benefits of mammography screening. The purpose of this study is to understand how objective risk information influences outcomes including behavioral intentions, attitudes about mammography, and emotional responses.

After participants view objective risk information, a post-test survey will measure outcome variables including behavioral intentions, knowledge, and emotional responses.

After reading information based on their condition, study participants will be asked to complete a series of questions to measure their reactions based on their condition. Specifically, the investigators will be measuring the following dependent variables (primary outcomes): behavioral intentions to receive mammograms, attitudes about mammography, subjective norms about mammography and breast cancer screening, knowledge about mammography outcomes and screening recommendations, and emotional responses to the material including psychological reactance. These outcomes will be measured using self-reported questionnaire items.

In this project, the investigators will compare alternative communication strategies to determine which strategy or strategies result in the greatest level of understanding. The investigators also will examine if the various strategies differentially affect the primary outcomes listed above.

ELIGIBILITY:
Inclusion Criteria:

* Adult women between the ages of 35 and 49 will be invited to participate in this study.

Exclusion Criteria:

* Women who have been previously diagnosed with breast cancer or have tested positive for the breast cancer gene will not be included.

Ages: 35 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1560 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12-18 (Actual); Study Completion 2012-12-18 (Actual)

PRIMARY OUTCOMES:
Behavioral intentions to get a mammogram | immediately following intervention (time 0)
  All participants will be asked to report their behavioral intentions to obtain mammograms in their 40s and at age 50.

SECONDARY OUTCOMES:
Attitude about mammography | immediately following intervention (time 0)
  Participants will be asked to report their attitudes about mammography (i.e., is a mammogram useful, harmful, etc.)

OTHER OUTCOMES:
Injunctive and descriptive norms about mammography | immediately following intervention (time 0)
  Participants will be asked to report their perceived norms about mammography, what they think important others would expect them to do and what they think other women their age or older are doing.
Decisional satisfaction | immediately following intervention (time 0)
  This variable assesses how satisfied participants feel about making a decision about mammography given the information they have been provided. Items include, "The information in the decision aid made me feel the choice to get a mammogram is being taken away from me by the groups that make screening recommendations."
Risk perception | immediately before and after intervention (time 0)
  This variable includes perceived severity and perceived susceptibility of breast cancer. Items include, "What is the chance that an average 40-49 year old woman will develop breast cancer in the next 10 years? Please choose a number between 0 (no chance of breast cancer) and 100 (definitely will get breast cancer)."
Clarity of the information being presented | immediately following intervention (time 0)
  These items assess how easy it is for participants to understand the numerical information that is provided in the decision aid.
Credibility of the information | immediately following intervention (time 0)
  These items measure the perceived trustworthiness, credibility, and accuracy of the information provided in the decision aid. Items include, "How credible did you find the information presented in the decision aid?"
Emotional reactions | immediately following intervention (time 0)
  The outcome includes measures of psychological reactance, anger, and fear that may be possible reactions to the decision aid. Items include, "How much do each of the following words (i.e., angry, worried) describe how you felt while reading the decision aid?"

CONTACTS AND LOCATIONS:
Overall Officials: Joseph N Cappella, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States